CLINICAL TRIAL: NCT06015360
Title: Using Fat Tissue GRafting to Treat Symptoms of VAginal Stenosis in Women With Gynaecological Cancer - IDEAL Stage 2a Surgical Study
Brief Title: Fat Grafting for Vaginal Stenosis in Gynaelogical Cancer
Acronym: GRASS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR5742
Record Dates: First submitted 2023-06-08; First posted 2023-08-29 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fat Grafting (Experimental): The fat grafting procedure will be conducted as per local standard RM protocol. All procedures will be conducted by the study Principal Investigator (PI) who is well practiced in performing this procedure in Head & Neck and breast cancer patients and also in scar revision patients.
  Interventions: Procedure: Fat Graft

INTERVENTIONS:
Procedure: Fat Graft — Fat grafting

SUMMARY:
The GRASS study looks at performing a technique called "Fat Tissue Grafting" to assess whether it can reduce the side effects of vaginal stenosis effects and improve the sexual function of participants who wish to preserve penetrative sexual function

DETAILED DESCRIPTION:
Vaginal stenosis is a common sequelae of radiotherapy treatment for cervical cancer. This can cause significant sexual problems resulting in sexual avoidance, relationship problems, feelings of low self-esteem, isolation, and difficulties initiating new relationships. Vaginal changes resulting in narrowing (stenosis) and adhesions can also lead to painful vaginal examinations which are routinely performed during follow-up consultations.

The available treatments for vaginal problems include regular use of vaginal dilators, lubricants, and moisturisers, all of which have shown poor results despite requiring an incessant effort by women.

A technique called 'fat grafting' has been successfully and safely used for many years to rectify the cosmetic and functional consequences of Breast and Head and Neck Cancers treatments. This technique is performed under general anaesthesia and uses fat tissue that is removed from other parts of the body; usually thighs, abdomen, and buttocks, by liposuction. The fat tissue is then processed into liquid and injected into the required area to generate more elasticity and improve tissue quality. To our knowledge this technique has never been applied to the field of Gynaecology-oncology.

In 2021 this technique was used in one patient with severe vaginal stenosis after radiotherapy treatment for advanced cervical cancer, by the Gynaecological and Plastic surgical teams at the Royal Marsden Hospital (RM). The fat tissue was harvested and processed using the method as described and injected into the vagina area (rectovaginal wall) with the aim being to generate more elasticity and improve the quality of the vaginal tissue. As a result of the procedure, the patient now reports reduction in vaginal bleeding and pain experienced, and a noticeable improvement in the size of the vagina allowing for penetrative sex.

This innovative technique addresses a neglected and unmet need of women to manage a consequence of curative treatment that is underreported and often unrecognised. It also serves as an example of how cross-discipline work focused on real patients' needs can produce ground-breaking solutions to complex clinical conundrums, by mobilising highly specialist clinical experts.

If this programme is successful, it can be expanded to women with vaginal stenosis due to radiotherapy for other cancers e.g., colorectal, or urological cancer. In addition, the investigators the investigators will work in partnership with the patient(s) who successfully benefit from fat grafting treatment to guide the development of a larger study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cervical cancer
* At least 2 years since finishing pelvic radiotherapy for gynaecological cancer
* Treated at RM
* Persistent symptoms of vaginal stenosis despite prior use of vaginal dilators/ oestrogen replacement / lubricants/moisturisers
* Desiring vaginal intercourse

Exclusion Criteria:

* Evidence of recurrent disease documented on Magnetic Resonance Imaging (MRI)
* Patients unwilling / unable to provide written informed consent for the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female patients
Enrollment: 8 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients able to have vaginal penetration without pain (yes / no) | 11 months
  Ability to have vaginal penetration , this is descriptive and will be provided as a yes / no answer by the patient at their follow up visit
Number of patients with an increase in the volume of the rectovaginal septum on pelvic MRI imaging | 10 months
  Increase in the volume of the rectovaginal septum on pelvic MRI imaging
Number of patients with reduced scarring on vaginal biopsies | 10 months
  Fat:Fibrosis ratio and total far and fibrosis percentage (as a percentage of the total stroma)
Improvement in sexual wellbeing | 11 months
  Measured using the Sexual Well-Being After Cervical or Endometrial Cancer (SWELL-CE) questionnaire (11) - a score drop below 9 (a score of 9 or above represents significant sexual difficulties)
Improvement in cervical cancer specific quality of life | 11 months
  Cervical cancer specific quality of life measured using the EORTC (European Organisation for Research and Treatment of Cancer) QLQ-CX24 - 10% improvement of the scale range for MCID (minimally clinically important differences)
Improvement in overall quality of life | 11 months
  Overall quality of life measured using the EORTC QLQ-C30. Any improvement in overall score will be deemed as an improvement
Improvement in overall quality of life | 11 months
  Overall quality of life measured using the EUROQOL EQ-5D-5L. Any improvement in overall score will be deemed as an improvement

SECONDARY OUTCOMES:
Occurrence of Calvien Dindo complications | 11 months
  Occurrence of Calvien Dindo complications (≥grade 3 ) post treatment
Determination of patient acceptability of the research procedure and of the trial | 11 months
  Determination of patient acceptability of the research procedure and of the trial will be explored in a focus group
Recruitment | 6 months
  Number of patients screened eligible, number approached and number of patients who consent to take part
Retention | 12 months
  Assess the proportion of patients who complete each planned fat graft treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No